CLINICAL TRIAL: NCT02844192
Title: Pharmacokinetics of Vancomycin in ICU Patients
Acronym: PK-VANCO-ICU
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0452
Record Dates: First submitted 2016-07-12; First posted 2016-07-26 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Suspected Infection With Vancomycin Susceptible Bacterial Strains
Keywords: Vancomycin; under dosage; intensive care unit; pharmacokinetics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Vancomycin is frequently under-dosed in ICU patients during the first 24-48 hours of treatment. Glomerular hyperfiltration syndrome, increased drug volume of distribution, vasopressor use, male sex and hypoalbuminemia are identified risk factor for vancomycin underdosing in ICU patients, among others.

To date, bedside estimation of vancomycin volume of distribution is challenging, and new methods for optimizing drug administration are required.

The Picco device is a moderately invasive hemodynamic monitoring system, providing parameters that may help estimation of vancomycin pharmacokinetics parameter.

The aim of this study is to test whether addition of hemodynamic parameters would improve pharmacokinetics modelling of vancomycin concentration in ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* patient hospitalized in intensive care unit
* under intravenous vancomycin started during current ICU hospitalization
* with at least one vancomycin serum concentration available
* under hemodynamic monitoring with the Picco ® device

Exclusion Criteria:

* vancomycin treatment for less than 24 hours
* vancomycin concentration in serum unavailable
* rare comorbidities influencing vancomycin pharmacokinetics

  * myeloma
  * cystic fibrosis
  * burn injury on more than 20 % of the body surface
* previous inclusion in present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-10; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Akaike information criterion as a measurement of goodness of fit of pharmacokinetic modeling of vancomycin serum concentration | week 1
  All available vancomycin measurements during the first week of treatment will be included in the pharmacokinetics model.
  All vancomycin dosages up to seven days of treatment will be used in a population pharmacokinetic model and an individual pharmacokinetic model

SECONDARY OUTCOMES:
Rate of patients with under-dosage of vancomycin at day 2 of treatment | day 2
  under-dosage of vancomycin is defined by a vancomycin serum concentration below 15 mg/l on day 2 of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe RICHARD, Prof, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon - Hôpital de la Croix-Rousse - Réanimation, Surveillance Continue Médicales et Assistance Respiratoire,103 Grande Rue de la Croix-Rousse, Lyon, France